CLINICAL TRIAL: NCT05746429
Title: Culturally Adapted Mobile Treatment of Chronic Pain in Adolescent Survivors of Pediatric Bone Sarcoma
Brief Title: Culturally Adapted Mobile Treatment of Chronic Pain in Adolescent Survivors of Pediatric Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ADAPTED; NCI-2022-10013 (Other: NCI Clinical Trial Registration Program); R61CA280978 (NIH)
Record Dates: First submitted 2023-01-10; First posted 2023-02-27 (Actual); Results first posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Bone Sarcoma; Childhood Cancer
MeSH Terms: conditions — Bone Neoplasms; Neoplasms | interventions — Cognitive Behavioral Therapy; Transcranial Direct Current Stimulation; Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Arm I (mobile CBT + active tDCS) (Experimental): Participants receive mobile CBT and undergo active tDCS to the dorsolateral prefrontal cortex (DLPFC) over 20 minutes twice a week for 6 weeks.
  Interventions: Behavioral: Cognitive Behavior Therapy; Device: Transcranial Direct Current Stimulation; Other: Questionnaire Administration
- Arm II (mobile CBT + sham tDCS) (Sham Comparator): Participants receive mobile CBT and undergo sham tDCS to the DLPFC over 20 minutes twice a week for 6 weeks.
  Interventions: Behavioral: Cognitive Behavior Therapy; Drug: Placebo Administration; Other: Questionnaire Administration
- Interview (Experimental): Participants attend virtual meetings and virtual focus groups during the cultural adaptation phase. Feedback is collected and analyzed to develop the finalized adaptation.
  Interventions: Other: Interview

INTERVENTIONS:
Behavioral: Cognitive Behavior Therapy — Receive mobile CBT
  Other Names: CBT, CBT, cognitive behavior therapy, cognitive therapy, CT
  Arms: Arm I (mobile CBT + active tDCS); Arm II (mobile CBT + sham tDCS)
Device: Transcranial Direct Current Stimulation — Undergo active tDCS
  Other Names: tDCS
  Arms: Arm I (mobile CBT + active tDCS)
Drug: Placebo Administration — Undergo sham tDCS
  Arms: Arm II (mobile CBT + sham tDCS)
Other: Questionnaire Administration — Ancillary studies
  Arms: Arm I (mobile CBT + active tDCS); Arm II (mobile CBT + sham tDCS)
Other: Interview — Attend virtual meetings and focus groups
  Arms: Interview

SUMMARY:
This is a prospective study that will conduct a series of focus groups with non-Hispanic Black and Hispanic childhood cancer survivors to obtain their input on culturally adapting a mobile CBT program for chronic pain and tDCS procedures. Once this adaptation process is completed, the investigators will conduct a feasibility trial with non-Hispanic Black, Hispanic and non-Hispanic White survivors of childhood cancer with chronic pain. The feasibility study will assign eligible participants to either culturally adapted mobile CBT + active tDCS to the dorsolateral prefrontal cortex or culturally adapted mobile CBT + sham tDCS. We anticipate approximately 60 participants for the focus groups and approximately 30 participants for the feasibility study for a total of about 90 participants.

DETAILED DESCRIPTION:
Survivors of pediatric childhood cancer are at-risk for developing chronic pain. Cognitive behavioral therapy (CBT) is an effective non-pharmacologic treatment for chronic pain, and can be delivered remotely to reduce access barriers. However, these programs have not been adapted to be culturally sensitive to underserved populations thus limiting their reach, usefulness, and uptake. The investigators propose to culturally tailor an established, evidence-based mobile CBT program for chronic pain to Black and Hispanic adolescent survivors of childhood cancer. Once the program is fully adapted, we propose to pair the culturally adapted mobile CBT program with remotely delivered transcranial direct current stimulation (tDCS), which may enhance pain control in survivors. The investigators will conduct a 6-week feasibility study in a racially/ethnically diverse sample of non-Hispanic White, non-Hispanic Black, and Hispanic adolescent survivors of pediatric childhood cance with chronic pain using culturally adapted CBT paired with remote tDCS. Study results will inform the development of a randomized clinical trial.

ELIGIBILITY:
Inclusions Criteria for cultural adaption

* Adult
* Hispanic or non-Hispanic Black childhood cancer survivor or parent of Hispanic or non-Hispanic Black childhood cancer survivor
* 18 years or older
* Adolescents
* 10-17 years-old survivors of childhood cancer
* At least one year post treatment
* Hispanic or non-Hispanic Black
* Phase 4 only: History of chronic pain (i.e. pain that was present for more than 3 months)

Exclusion Criteria for cultural adaptation

* Adults/Adolescents
* Inability or unwillingness of research participants or legal guardian/representative to give written informed consent

Inclusion Criteria for feasibility study

* Hispanic, non-Hispanic Black and non-Hispanic White 10-17-year-old survivors of pediatric cancer
* At least one year post treatment
* Pain present over the past 3 months and pain at least once per week
* Pain interfering with at least one area of daily functioning

Exclusion Criteria for feasibility study

* Limb amputation
* History of seizures or other neurological disorders
* Implanted medical device or metal in the head
* Serious comorbid psychiatric condition
* Current substance abuse
* History of development delay or significant cognitive impairment
* History of brain tumor diagnosis

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2023-04-06 (Actual); Primary Completion 2024-10-29 (Actual); Study Completion 2024-10-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tara Brinkman, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From April 2023 to August 2024, 68 participants were enrolled across two phases. Phase 1, a cultural adaptation study, included 38 participants in qualitative focus groups. Phase 2, a feasibility clinical trial with two arms, enrolled 33 participants. Three adolescents participated in both phases.
Pre-assignment Details: In the cultural adaptation phase, participants took part in focus groups and did not receive any intervention. In the feasibility study, all participants received the adapted mobile CBT. Participants were also assigned to active or sham transcranial direct current stimulation (tDCS) using an ABAB design within racial/ethnic groups (Hispanic, non-Hispanic Black, non-Hispanic White).
Groups:
- Experimental: Interview: Participants attend virtual meetings and virtual focus groups during the cultural adaptation phase. Feedback is collected and analyzed to develop the finalized adaptation.
- Experimental: Arm I (Mobile CBT + Active tDCS): Participants receive mobile CBT and undergo active tDCS to the DLPFC over 20 minutes twice a week for 6 weeks.
- Sham Comparator: Arm II (Mobile CBT + Sham tDCS): Participants receive mobile CBT and undergo sham tDCS to the DLPFC over 20 minutes twice a week for 6 weeks.
Period: Cultural Adaptation
Arm/Group | Experimental: Interview | Experimental: Arm I (Mobile CBT + Active tDCS) | Sham Comparator: Arm II (Mobile CBT + Sham tDCS)
Started | 38 | 0 | 0
Completed | 38 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Feasibility Study
Arm/Group | Experimental: Interview | Experimental: Arm I (Mobile CBT + Active tDCS) | Sham Comparator: Arm II (Mobile CBT + Sham tDCS)
Started | 0 | 15 | 18
Completed | 0 | 14 | 16
Not Completed | 0 | 1 | 2
Not completed — Lost to Follow-up | 0 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental: Interview | Experimental: Arm I (Mobile CBT + Active tDCS) | Sham Comparator: Arm II (Mobile CBT + Sham tDCS) | Total
Number analyzed (Participants) | 38 | 14 | 16 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.00 (14.12) | 14.69 (2.17) | 13.17 (2.18) | 20.10 (11.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 9 | 8 | 43
  Male | 12 | 5 | 8 | 25
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 20 | 5 | 5 | 30
  Non-Hispanic White | 0 | 5 | 6 | 11
  Hispanic or Latino | 18 | 4 | 5 | 27
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 38 | 14 | 16 | 68

OUTCOME MEASURES:

1. Primary Outcome: Pain Intensity
Description: Efficacy of mobile CBT paired with active versus sham tDCS on pain intensity in adolescent survivors with chronic pain. The Brief Pain Inventory-Short Form (BPI) includes a 4-item pain severity scale. Participants rate their worst and least pain in the last 24 hours, average pain, and current pain using a 10-point rating scale (0=no pain to 10=pain as bad as you can imagine). The pain severity score was calculated as the average of the 4 items, with scores ranging between 0 and 10. Higher scores indicate greater pain intensity. Changes in pain intensity from baseline (enrollment) up to 8 weeks from the start of the intervention in the active treatment and placebo groups were reported.
Time Frame: Baseline (enrollment) and up to 8 weeks from start of feasibility study
Population: Include participants in the feasibility study who were assigned to an experimental arm and completed both the baseline and 6-week assessment. All participants were included in the analysis.
Measure: Mean (Standard Deviation); unit: Change in scores on a scale
Arm/Group | Experimental: Arm I (Mobile CBT + Active tDCS) | Sham Comparator: Arm II (Mobile CBT + Sham tDCS)
Number analyzed (Participants) | 14 | 16
Change in scores on a scale | -0.96 (1.7) | -0.56 (2.5)

2. Primary Outcome: Pain Interference
Description: Efficacy of mobile CBT paired with active versus sham tDCS on pain interference in adolescent survivors with chronic pain. Using the BPI, participants rate the impact of pain on general activity, mood, walking ability, normal work/school, relationships with other people, sleep and enjoyment of life using a 10-point rating scale (0=does not interfere to 10=completely interferes). The pain interference score was calculated as the average of the 7 items, with scores ranging between 0 and 10. Higher scores indicate greater pain interference. Changes in pain interference from baseline (enrollment) up to 8 weeks from the start of the intervention in the active treatment and placebo groups were reported.
Time Frame: Baseline (enrollment) and up to 8 weeks from start of feasibility study
Population: Include participants in the feasibility study who were assigned to an experimental arm and completed the 6-week assessment. All participants were included in the analysis.
Measure: Mean (Standard Deviation); unit: Change in scores on a scale
Arm/Group | Experimental: Arm I (Mobile CBT + Active tDCS) | Sham Comparator: Arm II (Mobile CBT + Sham tDCS)
Number analyzed (Participants) | 14 | 16
Change in scores on a scale | -0.60 (1.66) | -1.30 (2.16)

3. Primary Outcome: Pain Catastrophizing
Description: The Pain Catastrophizing Scale, Child version (PCS-C) is a 13-item self-report measure of overly negative attitudes of pain. It consists of three scales of rumination, magnification and helplessness. The measure uses a 5-point rating scale (0=not at all true to 4=very true). The scores of three subscales were calculated as the sum of specific items: Rumination (4 items; score range 0-16), Magnification (3 items; score range 0-12), and Helplessness (6 items; score range 0-24). The total score was calculated as the sum of all 13 items (score range 0-52). Higher scores indicate worse outcomes (i.e., more pain rumination, magnification, helplessness and overall pain catastrophizing). Changes in pain catastrophizing from baseline (enrollment) up to 8 weeks from the start of the intervention in the active treatment and placebo groups were reported.
Time Frame: Baseline (enrollment) and up to 8 weeks from start of feasibility study
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Change in scores on a scale
Arm/Group | Experimental: Arm I (Mobile CBT + Active tDCS) | Sham Comparator: Arm II (Mobile CBT + Sham tDCS)
Number analyzed (Participants) | 14 | 16
Change in scores on a scale
  Rumination | -0.07 (3.95) | -1.13 (3.96)
  Magnification | -0.64 (4.31) | -0.69 (3.4)
  Helplessness | 1.07 (4.91) | -1.81 (5.27)
  Total score | 0.36 (10.69) | -3.63 (11.02)

4. Primary Outcome: Depression
Description: The Patient-Reported Outcomes Measurement Information (PROMIS) Pediatric Depressive Symptoms is an 8-item measure of self-reported symptoms of low mood in children and adolescents over the past 7 days. The measure has a 5-point rating scale (Never to Almost Always). The PROMIS Health Measures Scoring Service was used to convert raw scores to T-scores (population mean=50 and standard deviation=10. Higher scores indicate more severe depressive symptoms. Changes in depressive symptoms from baseline (enrollment) up to 8 weeks from the start of the intervention in the active treatment and placebo groups were reported.
Time Frame: Baseline (enrollment) and up to 8 weeks from start of feasibility study
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Change in T-scores
Arm/Group | Experimental: Arm I (Mobile CBT + Active tDCS) | Sham Comparator: Arm II (Mobile CBT + Sham tDCS)
Number analyzed (Participants) | 14 | 16
Change in T-scores | -0.65 (9.43) | -3.13 (13.30)

5. Primary Outcome: Anxiety
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS) Pediatric Anxiety is an 8-item measure of self-reported symptoms of anxiety symptoms in children and adolescents over the past 7 days. The measure has a 5-point rating scale (Never to Almost Always). The PROMIS Health Measures Scoring Service was used to convert raw scores to T-scores (population mean=50 and standard deviation=10). Higher scores indicate more severe anxiety symptoms. Changes in anxiety symptoms from baseline (enrollment) up to 8 weeks from the start of the intervention in the active treatment and placebo groups were reported.
Time Frame: Baseline (enrollment) and up to 8 weeks from start of feasibility study
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Change in T-scores
Arm/Group | Experimental: Arm I (Mobile CBT + Active tDCS) | Sham Comparator: Arm II (Mobile CBT + Sham tDCS)
Number analyzed (Participants) | 14 | 16
Change in T-scores | -3.82 (7.51) | -2.01 (10.36)

6. Primary Outcome: Cancer-related Worry
Description: The Fear of Cancer Recurrence Inventory is a 9-item measure developed specifically for survivors of childhood cancer (8-18 years) to assess the presence of fear of recurrence and perceived risk recurrence. The measure has 5-point rating scale (0=Not at All to 4=A Great Deal). The total score was calculated as the sum of all 9 items, with scores ranging between 0 and 36. Higher scores indicate greater cancer-related worry. Changes in cancer-related worry symptoms from baseline (enrollment) up to 8 weeks from the start of the intervention in the active treatment and placebo groups were reported.
Time Frame: Baseline (enrollment) and up to 8 weeks from start of feasibility study
Population: Include participants in the feasibility study who were assigned to an experimental arm and completed the 6-week assessment. One participant with incomplete data on the Fear of Cancer Recurrence Inventory was excluded from the analysis.
Measure: Mean (Standard Deviation); unit: Change in scores on a scale
Arm/Group | Experimental: Arm I (Mobile CBT + Active tDCS) | Sham Comparator: Arm II (Mobile CBT + Sham tDCS)
Number analyzed (Participants) | 14 | 15
Change in scores on a scale | 3.64 (5.69) | -4.13 (6.51)

7. Primary Outcome: Physical Functioning
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS) Pediatric Mobility is an 8-item measure of self-reported ability at physical activities in children and adolescents in the past 7 days. The PROMIS Pediatric Upper Extremity is an 8-item measure of self-upper extremity function in the past 7 days. Both measures have a 5-point rating scale (No Trouble to Not Able to Do). For both measures, the PROMIS Health Measures Scoring Service was used to convert raw scores to T-scores (population mean=50 and standard deviation=10). Higher scores indicate better outcomes (i.e., greater mobility and upper extremity function, respectively). Changes in physical functioning from baseline (enrollment) up to 8 weeks from the start of the intervention in the active treatment and placebo groups were reported.
Time Frame: Baseline (enrollment) and up to 8 weeks from start of feasibility study
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Change in T-scores
Arm/Group | Experimental: Arm I (Mobile CBT + Active tDCS) | Sham Comparator: Arm II (Mobile CBT + Sham tDCS)
Number analyzed (Participants) | 14 | 16
Change in T-scores
  Mobility | 0.34 (3.50) | 4.03 (9.47)
  Upper extremity | 1.94 (3.50) | 0.42 (6.48)

8. Primary Outcome: Peer Relations
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS) Pediatric Peer Relationship is an 8-item measure that assesses the quality of peer relationships. The measure has a 5-point rating scale (Never to Almost Always). The PROMIS Health Measures Scoring Service was used to convert raw scores to T-scores (population mean=50 and standard deviation=10). Higher scores indicate better quality relationships with peers. Changes in peer relationship quality from baseline (enrollment) up to 8 weeks from the start of the intervention in the active treatment and placebo groups were reported.
Time Frame: Baseline (enrollment) and up to 8 weeks from start of feasibility study
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Change in T-scores
Arm/Group | Experimental: Arm I (Mobile CBT + Active tDCS) | Sham Comparator: Arm II (Mobile CBT + Sham tDCS)
Number analyzed (Participants) | 14 | 16
Change in T-scores | -1.64 (5.92) | -3.26 (10.69)

9. Primary Outcome: Fatigue
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS) Pediatric Fatigue is a 10-item measure that assesses symptoms of fatigue in the past 7 days. The measure has a 5-point rating scale (Never to Almost Always). The PROMIS Health Measures Scoring Service was used to convert raw scores to T-scores (population mean=50 and standard deviation=10). Higher scores indicate more fatigue. Changes in fatigue from baseline (enrollment) up to 8 weeks from the start of the intervention in the active treatment and placebo groups were reported.
Time Frame: Baseline (enrollment) and up to 8 weeks from start of feasibility study
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Change in T-scores
Arm/Group | Experimental: Arm I (Mobile CBT + Active tDCS) | Sham Comparator: Arm II (Mobile CBT + Sham tDCS)
Number analyzed (Participants) | 14 | 16
Change in T-scores | -2.72 (9.92) | -2.86 (10.14)

10. Primary Outcome: Sleep (Adolescent Sleep Wake Scale (ASWS))
Description: The Adolescent Sleep Wake Scale (ASWS) short form is a 10-item measure of behavioral sleep patterns in adolescents. The measure has a 6-point rating scale (1=Never to 6=Always). The total score was calculated as the average of the 10 items, with scores ranging between 0 and 6. Higher scores indicating better success of sleep quality. Changes in sleep from baseline (enrollment) up to 8 weeks from the start of the intervention in the active treatment and placebo groups were reported.
Time Frame: Baseline (enrollment) and up to 8 weeks from start of feasibility study
Population: Include participants in the feasibility study who were assigned to an experimental arm and completed the 6-week assessment. One participant with incomplete data on the Adolescent Sleep Wake Scale (ASWS) short form was excluded from the analysis.
Measure: Mean (Standard Deviation); unit: Change in scores on a scale
Arm/Group | Experimental: Arm I (Mobile CBT + Active tDCS) | Sham Comparator: Arm II (Mobile CBT + Sham tDCS)
Number analyzed (Participants) | 14 | 15
Change in scores on a scale | -0.20 (0.96) | 0.61 (0.74)

11. Primary Outcome: Sleep (PROMIS Sleep-related Impairment)
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep-Related Impairment 8-item measure to allow for assessment of sleep quality during the night as well as the impact of sleepiness on daytime function. This measure assesses sleep-related impairment over the past 7 days. The measure has a 5-point rating scale (Never to Always). The PROMIS Health Measures Scoring Service was used to convert raw scores to T-scores (population mean=50 and standard deviation=10). Higher scores indicate more sleep problems. Changes in sleep from baseline (enrollment) up to 8 weeks from the start of the intervention in the active treatment and placebo groups were reported.
Time Frame: Baseline (enrollment) and up to 8 weeks from start of feasibility study
Population: Include participants in the feasibility study who were assigned to an experimental arm and completed the 6-week assessment. All participants were included in the analysis for the PROMIS Sleep-Related Impairment.
Measure: Mean (Standard Deviation); unit: Change in T-scores
Arm/Group | Experimental: Arm I (Mobile CBT + Active tDCS) | Sham Comparator: Arm II (Mobile CBT + Sham tDCS)
Number analyzed (Participants) | 14 | 16
Change in T-scores | -0.51 (6.58) | -2.76 (9.72)

12. Primary Outcome: Global Acceptability and Satisfaction With Treatment
Description: Acceptability and satisfaction with treatment will be assessed using a 5-point numerical rating scale (NRS) (strongly disagree to strongly agree). Higher score indicates greater acceptability and satisfaction. The answers were categorized as agree yes (strongly agree or agree) versus no (neither agree nor disagree, disagree, or strongly disagree).
Time Frame: Up to 8 weeks from start of feasibility study
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental: Arm I (Mobile CBT + Active tDCS) | Sham Comparator: Arm II (Mobile CBT + Sham tDCS)
Number analyzed (Participants) | 14 | 16
Participants
  Acceptable treatment: Yes (strongly agree or agree) | 3 | 10
  Acceptable treatment: No (neither agree or disagree, disagree, strongly disagree) | 11 | 6
  Positive experience with the treatment: Yes (strongly agree or agree) | 8 | 12
  Positive experience with the treatment: No (neither agree or disagree, disagree, strongly disagree) | 6 | 4

13. Primary Outcome: Opioid Use
Description: At each timepoint participants and/or their parents will be asked to list the names of their medications, doses taken, and the frequency with which the medications were taken over the past 2 weeks. Opioid doses will be converted to morphine equivalent doses (MED; in mg) using an opioid equivalence table. Changes in opioid use from baseline (enrollment) up to 8 weeks from the start of the intervention in the active treatment and placebo groups were reported.
  Note: no participants reported taking opioids during the study
Time Frame: Baseline (enrollment) and up to 8 weeks from start of feasibility study
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg-morphine equivalents (MME)
Arm/Group | Experimental: Arm I (Mobile CBT + Active tDCS) | Sham Comparator: Arm II (Mobile CBT + Sham tDCS)
Number analyzed (Participants) | 14 | 16
mg-morphine equivalents (MME) | 0 (0) | 0 (0)

14. Primary Outcome: Parental Depression
Description: Parental depression will be measured at each time point using the Patient Health Questionnaire 8-item (PHQ-8), a measure of symptoms of major depressive disorder. The Patient Health Questionnaire is a 4-point rating scale (0=Not at All to 3=Nearly Every Day). The total score was calculated as the sum of all 8 items, with scores ranging between 0 and 24. Higher scores indicate greater depression. . Changes in parental depression from baseline (enrollment) up to 8 weeks from the start of the intervention in the active treatment and placebo groups were reported.
Time Frame: Baseline (enrollment) and up to 8 weeks from start of feasibility study
Population: Include participants in the feasibility study who were assigned to an experimental arm and completed the 6-week assessment. One participant with incomplete data on the Patient Health Questionnaire 8-item (PHQ-8) was excluded from the analysis.
Measure: Mean (Standard Deviation); unit: Change in scores on a scale
Arm/Group | Experimental: Arm I (Mobile CBT + Active tDCS) | Sham Comparator: Arm II (Mobile CBT + Sham tDCS)
Number analyzed (Participants) | 13 | 16
Change in scores on a scale | -2.00 (2.52) | -1.19 (2.81)

15. Primary Outcome: Parental Anxiety
Description: Parental anxiety will be measured at each time point using the Generalized Anxiety Disorder 7-item (GAD-7), a measure of symptoms of generalized anxiety. The Generalized Anxiety Disorder measure is a 4-point rating scale (0=Not at 3=All to Nearly Every Day). The total score was calculated as the sum of all 7 items, with scores ranging between 0 and 21. Higher scores indicate greater anxiety. Changes in parental anxiety from baseline (enrollment) up to 8 weeks from the start of the intervention in the active treatment and placebo groups were reported.
Time Frame: Baseline (enrollment) and up to 8 weeks from start of feasibility study
Population: Include participants in the feasibility study who were assigned to an experimental arm and completed the 6-week assessment. Two participants with incomplete data on the Generalized Anxiety Disorder 7-item (GAD-7) were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: Change in scores on a scale
Arm/Group | Experimental: Arm I (Mobile CBT + Active tDCS) | Sham Comparator: Arm II (Mobile CBT + Sham tDCS)
Number analyzed (Participants) | 14 | 14
Change in scores on a scale | -0.93 (3.08) | -1.14 (2.35)

ADVERSE EVENTS:
Time Frame: In the cultural adaptation phase, adverse events were self-reported by participants at any point during the study phase, up to 2 months. In the feasibility study, adverse events based on current symptoms were surveyed prior to the first stimulation session and then twice per week, at the end of each stimulation session, for the 6 weeks of the intervention.
Description: In the cultural adaptation phase, adverse events were collected through non-systematic assessments.
  In the feasibility study, adverse events were systematically assessed. Adverse events were described as either tolerable or distressing by participants. If a participant reported an adverse event at the first stimulation session, any subsequent adverse event of the same intensity (tolerable or distressing) did not contribute towards the counting of new adverse events.
Arm/Group | Experimental: Interview | Experimental: Arm I (Mobile CBT + Active tDCS) | Sham Comparator: Arm II (Mobile CBT + Sham tDCS)
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/14 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/14 | 0/16
Other Adverse Events (participants affected / at risk) | 0/38 | 14/14 | 15/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental: Interview (N=38) | Experimental: Arm I (Mobile CBT + Active tDCS) (N=14) | Sham Comparator: Arm II (Mobile CBT + Sham tDCS) (N=16)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Increased perspiration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (12)
Itching (Skin and subcutaneous tissue disorders) | 0 (0) | 9 (47) | 9 (27)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Tingling (Skin and subcutaneous tissue disorders) | 0 (0) | 10 (60) | 14 (71)
Burning sensation (Skin and subcutaneous tissue disorders) | 0 (0) | 7 (21) | 7 (31)
Redness (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (13) | 3 (4)
Pain (Skin and subcutaneous tissue disorders) | 0 (0) | 6 (18) | 3 (7)
Headache (Nervous system disorders) | 0 (0) | 8 (19) | 7 (22)
Dizziness (Nervous system disorders) | 0 (0) | 2 (7) | 1 (3)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 2 (3) | 1 (1)
Ringing in ears (Ear and labyrinth disorders) | 0 (0) | 2 (7) | 3 (4)
Anxiety (General disorders) | 0 (0) | 0 (0) | 2 (2)
Poor concentration (General disorders) | 0 (0) | 5 (6) | 1 (6)
Restlessness (General disorders) | 0 (0) | 2 (2) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (2) | 1 (6)
Decreased energy (General disorders) | 0 (0) | 3 (4) | 2 (2)
Drowsiness (General disorders) | 0 (0) | 2 (2) | 2 (6)
Other (General disorders) | 0 (0) | 2 (2) | 3 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-04-02): https://cdn.clinicaltrials.gov/large-docs/29/NCT05746429/Prot_SAP_000.pdf
  • Informed Consent Form (2024-05-06): https://cdn.clinicaltrials.gov/large-docs/29/NCT05746429/ICF_001.pdf